CLINICAL TRIAL: NCT06332872
Title: Comparison Effectiveness of Oral Ivermectin , 1% Permethrin Shampoo and 4% Dimeticone Liquid Gel in the Treatment of Pediculosis Capitis Among School Children in Chachoengsao Province, Thailand
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M046q/66
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pediculus Capitis Infestation; Permethrin Adverse Reaction; Dimethicone Adverse Reaction; Permethrin Allergy; Dimethicone Allergy; Ivermectin; School-age Children
Keywords: Pediculosis capitis; head lice; pediculicides; School; Children; Permethrin; Shampoo; Ivermectin; Dimenticone; gel; liquid gel; pediculosis
MeSH Terms: conditions — Lice Infestations | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral ivermectin (Experimental): For the treatment of head lice infestation, participants are receiving two single doses of oral ivermectin on days 0 and 7 of the experiment. (spaced 7 days apart)
  Interventions: Drug: Oral Ivermectin
- Dimeticone liquid gel (Experimental): For the treatment of head lice infestation, participants are receiving one application of 4% dimenticone liquid gel on day 0 of the experiment.
  Interventions: Drug: 4% dimenticone liquid gel
- Permethrin shampoo (No Intervention): Participants are receiving two applications of 1% permethrin shampoo, which is the current drug of choice for Pediculosis capitis, on days 0 and 7. This group is defined as a control group.

INTERVENTIONS:
Drug: Oral Ivermectin — Oral formulation (3mg tablet) Dosage: 2 single doses of 200 mcg/kg given 7 days apart
  Arms: Oral ivermectin
Drug: 4% dimenticone liquid gel — topical formulation (liquid gel) only 1 application
  Arms: Dimeticone liquid gel

SUMMARY:
The goal of this clinical trial is to Comparison effectiveness of Oral ivermectin , 1% Permethrin shampoo and 4% Dimeticone liquid gel in the treatment of Pediculosis capitis, to assess the prevalence of lice and associated risk factors between severity groups by using questionnaire-based surveys and diagnostic tests among school children in Baan Nayao, Chachoengsao Province, Thailand.

The main questions it aims to answer are

* What is more effective between Oral ivermectin , 1% Permethrin shampoo and 4%Dimeticone liquid gel in the treatment of Pediculosis capitis in school children in Baan Nayao, Chachoengsao Province, Thailand?
* What is Prevalence and risk factors of being infected with in head lice in school and community?
* What is Side effects of Oral ivermectin , 1% Permethrin shampoo and 4%Dimeticone liquid gel?

Participants will receive three different drugs are

* oral ivermectin
* 4% Dimeticone liquid gel
* 1% Permethrin shampoo

Participants voluntarily received oral ivermectin as per medical prescription, with treatment outcomes, side effects, and satisfaction levels monitored following two treatment cycles. Those exhibiting persistent lice infestations were subsequently treated with 1% permethrin shampoo, the standard treatment, while alternatives were provided for individuals allergic to permethrin. These findings will contribute to formulating tailored, effective, and safe treatment regimens for future patients.

DETAILED DESCRIPTION:
Study design :

The study consists of two study designs: a quantitative study using a cross-sectional study to investigate the prevalence of head lice infestation and identify risk factors of head lice infestation among groups of population diagnosed with varying degrees of infestation; heavy, medium, and light. Additionally, a field trial will be conducted to compare the effectiveness of oral ivermectin, 1% Permethrin shampoo, and 4% Dimethicone liquid gel for treatment of Pediculosis capitis on days 0, 7, 14, and 28.

Study population :

The study population consists of students aged between 6 and 13 years old attending three schools located in Tha Kradan Subdistrict, Sanam Chai Khet District, Chachoengsao Province. The treatment allocation for head lice infestation is as follows: students at Na Yao border patrol police school will receive oral ivermectin, students at Ban Na Isan border patrol police school will receive 4% Dimethicone liquid gel, and students at Phu Ngam Wittaya School will receive 1% Permethrin shampoo. All volunteer groups must obtain consent by signing a parental consent form before participating in the project.

Sample size calculation :

Based on the previous study, Permethrin has an efficacy of 40%, while Ivermectin has an efficacy of 86.7%. By calculating the sample size using the formula for comparing proportions in two population groups, we obtain a sample size of 21 per group. To account for potential loss to follow-up or inability to contact participants, a 20% loss to follow-up rate is added, resulting in a final sample size of 26 individuals per group. Therefore, 78 individuals will be included in the data collection process.

Data collection :

Data collection was based on two questionnaires and data on head lice infection. The first questionnaire was a pre-treatment questionnaire asking for informed consent and a questionnaire regarding basic information. Factors that may be related to lice infection were the parents of the subjects who completed the questionnaire because the subjects were under 14 years of age. The second post-treatment questionnaire recorded information about allergic reactions. Potential adverse side effects of using the three groups of drugs and the number of lice from the second combing.

Data collection on lice infection in this study was based on methods from previous studies. Where lice infestation is defined as the presence of live lice. This is checked using a nit comb to check for live lice in the sunlight. Detection of nits with the ability to survive will also be considered positive. In this research Live lice can be checked by using a nit comb. The level of lice infection is divided into high levels. medium and little High levels of lice infestation means finding more than one lice after combing 1 time. Moderate lice infestation means finding lice after combing 1 time, an amount equal to 1 lice, and low level lice infestation means not found lice on the first attempt, but live lice or eggs were found after 20 rounds of combing and inspecting the area above the ears and below the neck. A nit comb was given to each participant to prevent lice from being infected through the head.

Protocol :

The data collection process began with the give a letter explaining information about the research and a request for informed consent document to participants. Those interested in participating in the research will go through a screening process for lice infection by the research team. The volunteer's identity was verified to match the code set by the researcher. Screening for history of drug allergies that volunteers in each group will receive. Along with informing volunteers and parents of how to give the medicine, including possible side effects and how to behave. In the first lice test, those diagnosed with lice were asked to complete a questionnaire about factors associated with lice infecting subjects with different levels of lice. Next, take oral ivermectin, wash your hair with 1% Permethrin shampoo and leave it for 10 minutes, or marinate your hair with 4% Dimeticone liquid gel and leave it for 15 minutes according to the school group that is divided. Then rinse off with clean water. Subsequently, follow-up was performed by screening for lice infection after drug use on days 0, 7, 14 and 28 of all samples. On day 7, results for all 3 groups were followed up and a second treatment was given in the Oral group. Ivermectin and 1% Permethrin shampoo are administered as the first dose. and follow up on the results of the treatment of lice in all 3 groups on the 14th and 28th day after receiving the first dose. The researcher will fill out a second questionnaire asking for information about allergies and side effects. Then the lice are scraped and a sample is collected and counted. Live lice, dead lice, and larval eggs Then the researcher will record all the numbers and information in the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. The participants are studying in Na Yao border patrol police school, Ban Na Isan border patrol police school or Phu Ngam wittaya school.
2. Approved consent from the participants' caretaker

Exclusion Criteria:

1. History of Allergic sensitization to these substances
2. The participants with chronic scalp disorder
3. Those who had used a pediculicide within the previous two weeks
4. Those who had recently used bleaches, dyes, or permanent wave products
5. Anyone taking trimethoprim or cotrimoxazole at evaluation or during the previous four weeks
6. Those who had participated in another clinical trial within one month

Additional exclusion criteria for ivermectin

1. Pregnancy
2. Body weight < 20 kg.
3. Loss to follow up in a second dose

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Comparison effectiveness of Oral ivermectin , 1% Permethrin shampoo and 4% Dimeticone liquid gel in the treatment of Pediculosis capitis | From enrollment to the end of treatment at 28 days
  Treatment of Pediculosis capitis was considered effective by the absence of live lice

SECONDARY OUTCOMES:
Prevalence of head louse infestation among school children in Chachoengsao Province, Thailand | From enrollment to the end of screening at 28 days
  Determined with a fine-toothed de-lousing comb to detect living head lice under natural sunlight by combing the hair 20 times in each portion of hair and visual observation above the ears and along the nape of the neck. The detection of viable nits (louse eggs) and nymphs is also considered positive.
Side effects of Oral ivermectin , 1% Permethrin shampoo and 4%Dimeticone liquid gel | From enrollment to the end of treatment at 28 days
  collected by post-treatment questionnaire about symptoms and allergic reactions after receive the treatment; oral Ivermectin, 4% Dimenticone liquid gel, or 1% Permethrin shampoo
The association factor of head lice infestation among school children in Chachoengsao Province, Thailand | From the enrollment to the end of treatment at 28 days
  Collected by pre-treatment questionnaire about factors that may be related to lice infection. The parents of the subjects will complete the questionnaire because the subjects were under 14 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Phramongkutklao college of medicine, Bangkok, Thailand